CLINICAL TRIAL: NCT01189344
Title: Levothyroxine Absorption in Morbidly Obese Patients Before and After Roux-en-Y Bariatric Surgery
Brief Title: Levothyroxine (L-T4) Absorption After Bariatric Surgery
Acronym: RYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Geraldo Medeiros-Neto, University of São Paulo Medical School
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1039/07
Record Dates: First submitted 2010-08-23; First posted 2010-08-26 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2007-06

CONDITIONS: Morbid Obesity
Keywords: Obesity; LT4; Absorption; Thyroid function
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Not surgical group (Experimental): The Nos surgical (NS) group includes 15 patients for whom bariatric surgery is planned. Body mass index (BMI) of this group of patients is ≥40 Kg/m2.
  Interventions: Drug: Levothyroxine
- Surgical group (Experimental): The Surgical (S) group includes 15 patients who had undergone Roux-en-Y bariatric surgery 2 to 3 months before inclusion in the study
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — 600 µg of oral levothyroxine(LT4. Blood samples were collected before and after LT4 administration

SUMMARY:
Intestinal absorption of levothyroxine (LT4) tablets depends on its dissolution in gastric acid secretion, which is reduced after bariatric interventions. Impaired LT4 absorption due to low gastric dissolution has been reported in patients with atrophic or chronic gastritis. The objective of this study is to evaluate the absorption of LT4 tablets in morbidly obese patients before and after Roux-en-Y bariatric surgery.

DETAILED DESCRIPTION:
LEVOTHYROXINE ABSORPTION IN MORBIDLY OBESE PATIENTS BEFORE AND AFTER ROUX-EN-Y BARIATRIC SURGERY INTRODUCTION Levothyroxine sodium (LT4) is an effective drug prescribed as replacement therapy for patients with hypothyroidism, as a controversial suppressive therapy for nodular thyroid disease and after surgical removal of thyroid cancer. Incidence rates of differentiated thyroid cancer of all sizes have increased both in men and women, as have the rates of autoimmune thyroiditis disease. It is estimated that 3.7% of the United States population has hypothyroidism, indicating that millions of people are in continuous use of LT4.

Absorption of LT4 formulations approximates 80% of the oral dose. It is reduced when LT4 is ingested concomitantly with several drugs including aluminum hydroxide, cholestyramine, sucralfate, ferrous sulphate, calcium carbonate, sodium polystyrene sulfonate, as well as with coffee and fiber supplements.

Intestinal absorption of LT4 depends primarily on its dissolution in gastric acid secretion. Therefore, may be affected by H. pylori infection and autoimmune gastritis. There are substantial interindividual variations in LT4 requirements dependent on patients age, gender and body size, with lean body mass being the major determinant of dose correction for LT4. Morbidly obese patients apparently have impaired LT4 absorption.

The prevalence of obesity has increased to epidemic proportions. Effective treatment may be achieved by bariatric surgeries, but these procedures are associated with several morbidities, such as gastrointestinal and nutritional complications. It is plausible to hypothesize that since bariatric interventions (such as Roux-en-Y) reduce gastric hydrochloric acid secretion, they may impair LT4 absorption.

OBJECTIVE The aim of this study was to evaluate the absorption of LT4 tablets in morbidly obese patients before and after bariatric surgery in order to determine the need for adjustment of LT4 doses.

MATERIAL AND METHODS

Patients Patients will be recruited from the Gastric Surgery Division of Hospital das Clínicas. Thirty morbidly obese patients will be divided in two groups. The NS group will include 15 patients for whom bariatric surgery is planned. Body mass index (BMI) of this group of patients has to be ≥40 Kg/m2. The S group will include 15 patients who had undergone Roux-en-Y bariatric surgery 2 to 3 months before inclusion in the study.

Clinical data and medication information were collected before recruitment. Exclusion criteria includes a previous diagnosis of thyroid cancer, diabetes mellitus in use of insulin, chronic or atrophic gastritis, and use of medications associated with impaired LT4 absorption.

All patients will signed an informed consent. The study was approved by the Ethical Committee of Hospital das Clínicas, University of São Paulo Medical School (CAPPesq N0 1039/07).

Methods Absorption of LT4 will be measured using a previously described nonisotopic method. After an overnight fast, a forearm intravenous catheter is inserted and two blood samples will be collected with a 30-minute interval before administration of 600 µg of oral LT4. Blood samples will be collected 30, 60, 120, 180, 240, 300, and 1440 minutes (24 hours) after administration of LT4. Patients will fast for five hours after receiving the drug. They will be then instructed to have a light meal in the evening and to return the next morning in a fasting state to collect the 24 hour sample.

Serum free T4 (FT4), total T4 (TT4) and serum TSH will be determined in all samples by electrochemiluminescence immunoassay (Roche Corporation, Indianapolis, IN, USA). The concentration of each hormone at baseline will be calculated as a mean of the two samples collected before the LT4 dose. To correct for endogenous hormone synthesis, the incremental rise of each hormone concentration (deltaTT4, deltaFT4, deltaTSH) will be calculated by subtracting the basal value from the subsequent time intervals samples. To evaluate LT4 absorption, the area under the curve of deltaTT4 and deltaFT4 from baseline to 240 minutes and to 300 minutes (AUC240, AUC300) as well as the peak of deltaTT4 and deltaFT4 concentrations will be determined.

Serum leptin will be measured by Human Leptin Elisa Kit (Millipore, Billerica, MA) in all patients, before and after weight loss following the surgery.

Chronic autoimmune gastritis will be ruled out by absence of clinical signs and negative antiparietal autoantibodies.

Statistical analysis Results will be expressed as mean±standard deviation (SD). Analysis of variance and Tukey Multiple Comparison test, Student's t test and Spearman correlation analysis will be performed to compare the data. All tests will be performed with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese individual (body mass index (BMI)≥40 Kg/m2)
* individuals for whom bariatric surgery is indicated
* patients who had undergone Roux-en-Y bariatric surgery 2 to 3 months before inclusion in the study

Exclusion Criteria:

* previous diagnosis of thyroid cancer
* diabetes mellitus in use of insulin
* chronic or atrophic gastritis
* use of medications associated with impaired LT4 absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Sherman SI, Malecha SE. Absorption and Malabsorption of Levothyroxine Sodium. Am J Ther. 1995 Oct;2(10):814-818. doi: 10.1097/00045391-199510000-00014. No abstract available. PMID 11854792